## The GlaxoSmithKline group of companies

| Division | · | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for an open-label study in healthy male subjects, to determine the excretion balance as pharmacokinetics of [14C]-GSK2269557, administered as a single intravenous microtracer (concomitant with an inhale non-radiolabelled dose) and a single oral dose |
|---|---|---|
| <b>Compound Number</b> | : | GSK2269557 |
| <b>Effective Date</b> | : | 09-JAN-2018 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206764.
- This RAP is intended to describe the safety and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## **RAP Author(s):**

| Approver | |
|---------------|-----------------------------|
| PPD | |
| Study Statist | ician (Clinical Statistics) |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Data Manager (Data Management) | 03-JAN-2018 | email |
| Manager (Clinical Pharmacology) | 05-JAN-2018 | email |
| Clinical Research Scientist (Clinical Sciences) | 04-JAN-2018 | email |
| Clinical Development Scientist (Clinical Development) | 04-JAN-2018 | email |
| Clinical Development Director (Clinical Development) | 03-JAN-2018 | email |
| Manager (Clinical Programming) | 08-JAN-2018 | email |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|--------------------------------|-------------|-----------------|
| Director (Clinical Statistics) | 09-JAN-2018 | email |
| Manager (Clinical Programming) | 09-JAN-2018 | email |

## **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | N | | 5 |
| 2. | SLIMA | /ΔRV ∩F | KEV PROT | FOCOL INFORMATION | 5 |
| ۷. | 2.1. | | | tocol Defined Statistical Analysis Plan | |
| | 2.1. | | | and Endpoint(s) | |
| | 2.3. | | | | |
| | 2.4. | Statistica | al Hynothes | ses / Statistical Analyses | 7 |
| | ۷.٦. | Otationo | arriypoulos | oco / Otaliolical Arialyses | |
| 3. | PLAN | NED ANA | LYSES | | 8 |
| | 3.1. | Final Ana | alyses | | 8 |
| | | | • | | |
| 4. | ANAL | | | S | |
| | 4.1. | Protocol | Deviations | i | 8 |
| 5. | | | | DATA ANALYSES AND DATA HANDLING | 40 |
| | | | | Cub are a Diagle Descriptor | |
| | 5.1.<br>5.2. | | | Sub-group Display Descriptors | |
| | 5.2.<br>5.3. | | | sns for Data Analyses and Data Handling | 10 |
| | 5.5. | | | Data Arialyses and Data Hariding | 10 |
| | | Convent | 10113 | | 10 |
| 6. | STUD | Y POPUL | ATION AN | ALYSES | 12 |
| - | 6.1. | | | ed Study Population Analyses | |
| 7. | SAFE | TY ANAL | YSES | | 13 |
| | 7.1. | | | alyses | |
| | 7.2. | | | Special Interest Analyses | |
| | 7.3. | | • | Analyses | |
| | 7.4. | Other Sa | afety Analys | ses | 13 |
| 8. | ДЦΛГ | | | ALYSES | 1.1 |
| Ο. | 8.1. | | _ | S | |
| | 0.1. | 8.1.1. | | centration Measures | |
| | | 8.1.2. | | Pharmacokinetic Parameters | |
| | 8.2. | - | | kinetic Analyses | |
| | 0.2. | 8.2.1. | | / Variables | |
| | | 0.2.1. | 8.2.1.1. | Drug Concentration Measures | |
| | | | 8.2.1.2. | Derived Pharmacokinetic Parameters | |
| | | 8.2.2. | • | Measure | |
| | | 8.2.3. | | n of Interest | |
| | | 8.2.4. | | Analyses / Methods | |
| | 8.3. | - | | cokinetic Analyses | |
| | | 8.3.1. | | / Variables | |
| | | | 8.3.1.1. | Drug Concentration Measures | |
| | | | 8.3.1.2. | Derived Pharmacokinetic Parameters | |
| | | 8.3.2. | Summary | Measure | <mark>21</mark> |
| | | 8.3.3. | | n of Interest | |
| | | 8.3.4. | Statistical | Analyses / Methods | 21 |

## CONFIDENTIAL

| $\sim$ | ე6 | 7/ | • |
|--------|----|-----|----|
| | ın | / r | ٦Δ |

| | | | 8.3.4.1. | Statistical Methodology Specification | 21 |
|---|---|---|---|---|---|
| 9. | EXPLO | ORATORY | / ANALYSE | :S | 23 |
| 10. | REFE | RENCES. | | | 24 |
| | A DDEA | IDIOEO | | | 0.5 |
| 11. | | | | I Deviation Management | |
| | 11.1.<br>11.2. | | | I Deviation Managementle of Activities | |
| | 11.2. | 11 2 1 | Protocol D | efined Schedule of Events | 20 |
| | 11.3. | | | Phases and Treatment Emergent Adverse | 20 |
| | 11.0. | | | | 30 |
| | | 11.3.1. | | ses | |
| | | 11.0.1. | | Study Phases for Concomitant Medication | |
| | | 11.3.2. | | Emergent Flag for Adverse Events | |
| | 11.4. | | | splay Standards & Handling Conventions | |
| | | 11.4.1. | | Process | |
| | | 11.4.2. | | Standards | |
| | | 11.4.3. | | Standards for Pharmacokinetic | |
| | 11.5. | Appendix | 5: Derived | and Transformed Data | 34 |
| | | 11.5.1. | | | |
| | | 11.5.2. | | ulation | |
| | | 11.5.3. | | | |
| | 11.6. | | | ng Standards for Missing Data | |
| | | 11.6.1. | | Withdrawals | |
| | | 11.6.2. | | f Missing Data | |
| | 44 7 | A | 11.6.2.1. | Handling of Missing and Partial Dates | 36 |
| | 11.7. | | | of Potential Clinical Importance | |
| | | 11.7.1. | | Values | |
| | | 11.7.2. | | | |
| | 11.8. | | Vilai Siyiis<br>V 8: Abbrevi | ations & Trade Marks | 38 |
| | 11.0. | 11.8.1. | | ons | |
| | | 11.8.2. | | (S | |
| | 11.9. | _ | | Data Displays | |
| | 11.0. | | | ay Numbering | |
| | | 11.9.2. | Mock Exar | nple Shell Referencing | .42 |
| | | 11.9.3. | | es | |
| | | 11.9.4. | | ulation Tables | |
| | | 11.9.5. | | kinetic Tables | |
| | | 11.9.6. | | kinetic Figures | |
| | | 11.9.7. | | oles | |
| | | 11.9.8. | _ | js | |
| | | 11.9.9. | | istings | |
| | 11.10. | Appendix | د 10: Examp | ole Mock Shells for Data Displays | 63 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2017N324843_00 | 09-AUG-2017 | Original |
| 2017N324843_01 | 30-OCT-2017 | Protocol Amendment 1 was put in place to: |
| | | <ul> <li>Respond to comments from the Regulatory Authority:<br/>Medicines and Healthcare Products Regulatory<br/>Authoring.</li> </ul> |
| | | <ul> <li>Reflect an update to the Investigator's Brochure (IB)<br/>published since approval of the original protocol.</li> </ul> |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 1 [(Dated: 30/Oct/2017)], however additional PK parameters have been requested.

## 2.2. Study Objective(s) and Endpoint(s)

| Objective | Endpoint |
|---|---|
| Primary | |
| To determine total radioactivity (drug related material) in plasma following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled GSK2269557 dose) and a single oral dose of [14C]-GSK2269557. | AUC (0-inf), AUC (0-t), Cmax, tmax, t1/2 of total drug-related material (radioactivity) in plasma. |
| To determine the rate and extent of excretion of total radioactivity in urine and faeces and the total recovery of radioactivity following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C]-GSK2269557. | Urinary and faecal cumulative excretion as<br>a percentage of the total radioactive dose<br>administered over time. |

| Objective | Endpoint |
|---|---|
| Seco | ndary |
| To determine parent GSK2269557 concentration in plasma following a single IV microtracer of [14C]-GSK2269557 concomitant with an inhaled non- radiolabelled GSK2269557 dose and a single oral dose of [14C]-GSK2269557. | <ul> <li>AUC(0-inf), AUC(0-t), Cmax, tmax, and t1/2 of parent GSK2269557 and [¹⁴C]-GSK2269557¹ in plasma.</li> <li>Volume and clearance of parent [¹⁴C]-GSK2269557¹ after IV dose only.</li> </ul> |
| To estimate the absolute bioavailability of GSK2269557 following inhaled and oral administration. | Oral and inhaled F (absolute bioavailability). |
| To evaluate the safety and tolerability of<br>GSK2269557 after single IV, oral and<br>inhaled doses in healthy participants. | <ul> <li>Incidence of adverse events.</li> <li>Laboratory safety, electrocardiogram (ECG) and vital signs parameters.</li> </ul> |
| Explo | ratory |
| To generate samples that will be used to characterise the metabolic profile of GSK2269557 in plasma, urine, faeces, and duodenal bile (following IV dose only), following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C]-GSK2269557 (these analytical investigations will be conducted and the results reported under a separate Platform Technology Services (PTS) In vitro/In vivo Translation (IVIVT), GlaxoSmithKline protocol). | Characterisation and quantification of metabolites in plasma, urine, faeces, and duodenal bile (these analytical investigations will be conducted and the results reported in a separate GSK PTS IVIVT protocol). |

<sup>1.</sup> For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by liquid chromatography (LC) + Accelerator Mass Spectrometry (AMS), whereas GSK2269557 describes the parent GSK2269557 concentration derived via liquid chromatography-tandem mass spectrometry (LC/MS).

Note: the above table is as presented in the protocol amendment, subsequently additional PK parameters have been requested including: plasma AUC(0-24) and %AUCex for parent GSK2269557 and total radioactivity analytes; plasma ML(iv), ML(po), Fg, EH, Fabs; parent GSK2269557/ total radioactivity ratios for the plasma PK parameters Cmax, AUC(0-t), AUC(0-24) and AUC(0- $\infty$ ); and CLr derivations are described in Section 8.

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

• No formal hypotheses will be tested or treatment comparisons performed. Data will be summarised using descriptive methods only.

## 3. PLANNED ANALYSES

## 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management. Note: pharmacokinetic concentration and pharmacokinetic parameter raw file generation start after GSK DBF take approx. 18 working days after DBF. All other datasets available at DBF.

## 4. ANALYSIS POPULATIONS

| Population | ppulation Definition / Criteria | |
|---|---|---|
| All Participants<br>Enrolled (APE)<br>Population | All participants for whom a record exists on the study database; includes both screened participants and participants who are not screened but sign the informed consent form (ICF). | Screen Failure |
| Safety Population | <ul> <li>Participants in the APE Population who receive at least one dose of study treatment.</li> <li>Participants will be analysed according to the treatment they actually received</li> </ul> | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) Population | <ul> <li>Participants in the APE Population who receive at least one dose of study treatment and for whom a PK sample was obtained and analysed.</li> <li>Participants will be analysed according to the treatment they actually received</li> </ul> | • PK |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

#### **CONFIDENTIAL**

206764

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the pCRF.

The study endpoints will be reported using the populations detailed in Section 4 of this document regardless of whether the subjects deviate from the protocol.

If there are subjects with protocol deviations that may potentially impact the PK endpoints, exploratory sensitivity summaries may be considered. If further summaries of the data are produced, they will be detailed in the clinical study report.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Data Displays for Reporting [1] | | | |
| Code | Description | Description | Order [2] |
| А | GSK2269557 1000 mcg Inhaled + [14C]-GSK2269557 10 mcg IV | 557 IH + 14C-557 IV | 1 |
| В | [14C]-GSK2269557 800 mcg Oral | 14C-557 ORAL | 2 |

#### NOTES:

- The following footnote will be presented on each display:
   557 IH + 14C-557 IV = Intravenous radiolabelled 10 mcg GSK2269557 co-administered with inhaled 1000 mcg GSK2269557; 14C-557 ORAL = 800 mcg radiolabelled GSK2269557 administered orally
- 2. Order represents treatments being presented in TFL, as appropriate

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Baseline definitions defined in the table are applicable to each "period" for this crossover study.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | Safety | | | |
| 12-Lead ECG | X | Χ | X | Day 1 (Pre Dose) |
| Vital Signs | X | Χ | X | Day 1 (Pre Dose) |
| Haematology | X | Х | Х | Day 1 (Pre Dose) |
| Clinical Chemistry | X | Χ | X | Day 1 (Pre Dose) |
| Liver Function | X | Χ | X | Day 1 (Pre Dose) |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing. The mean of triplicate measurements at any given time point will be used as the value for that time point unless otherwise stated.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

## **CONFIDENTIAL**

## 

| Section | Component |
|---------|---------------------------------------------------------------|
| 11.3 | Appendix 3 Study Phases and Treatment Emergent Adverse Events |
| 11.4 | Appendix 4 Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5 Derived and Transformed Data |
| 11.6 | Appendix 6 Reporting Standards for Missing Data |
| 11.7 | Appendix 7 Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9 List of Data Displays.

## 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9 List of Data Displays.

## 7.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. The details of the planned displays are provided in Appendix 9 List of Data Displays.

## 7.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9 List of Data Displays.

## 7.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9 List of Data Displays.

## 8. PHARMACOKINETIC ANALYSES

The plasma pharmacokinetic concentrations will have different nomenclatures dependent on the method of measuring. For measured concentrations of GSK2269557 in blood plasma, the nomenclature [14C]-GSK2269557 describes the parent GSK2269557 concentration derived via analysis by liquid chromatography (LC) + Accelerator Mass Spectrometry (AMS), whereas GSK2269557 describes the parent GSK2269557 concentration derived via liquid chromatography-tandem mass spectrometry (LC/MS). It is expected that, for period 1, the radiolabelled iv dose will be measured using LC+AMS and will be labelled "[14C]-GSK2269557", the non-radiolabelled inhaled dose will be measured using LC/MS and will be labelled "GSK2269557". For period 2, the radiolabelled oral dose will be measured using LC/MS and will be labelled "GSK2269557". For each period the total radioactivity will be measured by AMS and will be labelled "Total Radioactivity". However, these methods may be adapted if necessary.

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of, Clinical Pharmacology Science and Study Operations (CPSSO), GlaxoSmithKline.

Derivation of plasma pharmacokinetic parameters for [<sup>14</sup>C]-GSK2269557, total radioactivity and GSK2269557 will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

Derivation of urine/faeces total radioactivity parameters will be performed by, or under the direct auspices of Bioanalysis, Immunogenicity and Biomarkers (BIB), PTS IVIVT, GlaxoSmithKline.

## 8.1. Endpoint / Variables

#### 8.1.1. Drug Concentration Measures

Refer to Appendix 4 Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times.

Pharmacokinetic parameters listed in Table 1 will be determined from the plasma concentration-time data, as data permits, for each subject, analyte (total radioactivity, GSK2269557 and [<sup>14</sup>C]-GSK2269557) and treatment period unless otherwise stated.

Pharmacokinetic parameters listed in Table 2 will be determined from the urine and faeces concentration-time data, as data permits, for each collection interval, subject and treatment period unless otherwise stated.

 Table 1
 Derived Plasma Pharmacokinetic Parameters

| Parameter Description |
|---|
| Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Area under the concentration-time curve from time zero to 24 hours post dose (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| The percentage of AUC (0-∞) obtained by extrapolation (%AUCex) will be calculated as: |
| [AUC(0-inf) - AUC(0-t)] / AUC(0-inf) x 100 |
| Maximum observed concentration, determined directly from the concentration-time data. |
| Time to reach Cmax, determined directly from the concentration-time data. |
| Apparent terminal half-life will be calculated as: t½ = In2 / lambda_z |
| Total iv clearance will be calculated as: |
| CL(iv)=Dose(iv)/AUC(0-∞) |
| Treatment period 1, analyte [ $^{14}$ C]-GSK2269557 only where Dose(iv) is the actual iv dose calculated as [weight of full syringe (g) minus syringe weight after dose (g)] multiplied by nominal concentration ( $\mu$ g/g) |
| If Plasma AUC(0-∞) is calculable then CLr= Cumulative Ae[urine] for treatment period 1/Plasma AUC(0-∞) |
| If Plasma AUC(0-∞) is not calculable then CLr= Cumulative Ae[urine] for treatment period 1/Plasma AUC(0-t) |
| Where cumulative Ae from excretion data for treatment period 1 and AUC from NCA PK analysis of Treatment period 1, analyte [14C]-GSK2269557 only. |
| Dose(IV)/AUC(0-∞) |
| Treatment period 1, analyte [14C]-GSK2269557 only. |
| Where Dose(IV) is the radiometric dose as described in Table 1. |
| $Dose(IV) \times AUMC(0-\infty)/(AUC(0-\infty))^{2}$ |
| Treatment period 1, analyte [¹4C]-GSK2269557 only. |
| Where AUMC is the area under the moment curve and Dose(IV) is the radiometric dose as described in Table 1. |

| Parameter | Parameter Description |
|---|---|
| ML(iv) | Metabolite load following intravenous administration is calculated as: |
| | Total Radioactivity AUC(0-∞) – [14C]-GSK2269557 AUC(0-∞) |
| | Total Radioactivity AUC(0-∞) |
| | Treatment period 1 only |
| ML(po) | Metabolite load following oral administration is calculated as: |
| | Total Radioactivity AUC(0-∞) — GSK2269557 AUC(0-∞) |
| | Total Radioactivity AUC(0-∞) |
| | Treatment period 2 only. |
| | Note: GSK2269557 AUC(0-∞) may be updated depending on the sample analysis conducted but refers to the parent GSK2269557 from oral dose. |
| Fg | Fraction metabolised by gut wall as a fraction of the oral dose will be calculated as follows: |
| | Fg= 1 –(ML(po)–ML(iv)) |
| Ен | Hepatic extraction ratio is calculated (Davis, B et al, 1993) as follows: |
| | $E_{\rm H}$ = CL(iv)/1450 mL/min |
| F <sub>abs</sub> | Fraction absorbed following an oral dose is calculated as follows: |
| | $F_{abs} = \frac{\frac{\text{Oral } F(0-\infty)}{1-E_H}}{F_g}$ |
| Dose(IV) | Radiometric IV dose will be calculated by Covance |
| Dose(oral) | Radiometric Oral dose will be calculated by Covance |
| Dose(inhaled) | Nominal inhaled dose |
| Oral F (0-∞) | Oral absolute bioavailability based on AUC(0-∞) calculated as: |
| | $\frac{\text{GSK2269557 AUC}(0-\infty)(\text{oral})}{\text{Dose}(\text{oral})} / \underbrace{\frac{[14C]\text{-GSK2269557 AUC}(0-\infty)(\text{iv})}{\text{Dose}(\text{iv})}}$ |
| | Per subject. |
| | Note: Radiometric dose will be used for oral and iv as described in Table 1. GSK2269557 AUC(0-∞)(oral) may be updated depending on the sample analysis |

| Parameter | Parameter Description |
|---|---|
| | conducted but refers to the parent GSK2269557 from oral dose. |
| Inhaled F (0-∞) | Inhaled absolute bioavailability based on AUC(0-∞) calculated as |
| | GSK2269557 AUC(0-∞)(inhaled) , |
| | Dose(inhaled) |
| | /[14C]-GSK2269557 AUC(0-∞)(iv) Dose(iv) |
| | Per subject. |
| | Note: Radiometric dose will be used for oral and iv as described in Table 1. |
| Oral F (0-t) | Oral absolute bioavailability based on AUC(0-t) calculated as: |
| | GSK2269557 AUC(0-t)(oral) / |
| | Dose(oral) |
| | /[14C]-GSK2269557 AUC(0-t)(iv) Dose(iv) |
| | Per subject. |
| | Note: Radiometric dose will be used for oral and iv as described in Table 1 GSK2269557 AUC(0-∞)(oral) may be updated depending on the sample analysis |
| | conducted but refers to the parent GSK2269557 from oral dose. |
| Inhaled F (0-t) | Inhaled absolute bioavailability based on AUC(0-t) calculated as |
| | GSK2269557 AUC(0-t)(oral) / |
| | Dose(oral) /[14C]-GSK2269557 AUC(0-t)(iv) |
| | $ / \frac{[14C]\text{-GSK2269557 AUC(0-t)(iv)}}{\text{Dose(iv)}} $ |
| | Per subject. |
| | Note: Radiometric dose will be used for oral and iv as described in Table 1. |
| GSK2269557 | Cmax Ratio = Exp { [loge(GSK2269557 Cmax] - [loge(Total radioactivity Cmax]} |
| /Total radioactivity ratio for Cmax, | Per subject for radiolabelled oral dose. GSK2269557 may be updated depending on the sample analysis conducted but refers to the parent GSK2269557 from oral dose |
| GSK2269557 /Total radioactivity | AUC(0-inf) Ratio = Exp { [loge(GSK2269557 AUC(0-inf)] - [loge(Total radioactivity AUC(0-inf)] } |
| ratio for AUC(0-inf) | Per subject for radiolabelled oral dose. GSK2269557 may be updated depending on the sample analysis conducted but refers to the parent GSK2269557 from oral dose |
| GSK2269557 | AUC(0-t) Ratio = Exp { [loge(GSK2269557 AUC(0-t)] - [loge(Total radioactivity AUC(0- |
| /Total radioactivity | t)] } |

| Parameter | Parameter Description |
|---|---|
| ratio for AUC(0-t) | Per subject for radiolabelled oral dose. GSK2269557 may be updated depending on the sample analysis conducted but refers to the parent GSK2269557 from oral dose |
| [¹4C]-GSK2269557<br>/Total radioactivity<br>ratio for Cmax, | Cmax Ratio = Exp { [loge([14C]-GSK2269557 Cmax] - [loge(Total radioactivity Cmax]} Per subject for radiolabelled IV dose. |
| [¹4C]-GSK2269557<br>/Total radioactivity<br>ratio for AUC(0-inf) | AUC(0-inf) Ratio = Exp { [loge([14C]-GSK2269557 AUC(0-inf)] - [loge(Total radioactivity AUC(0-inf)] } Per subject for radiolabelled IV dose. |
| [¹⁴C]-GSK2269557<br>/Total radioactivity<br>ratio for AUC(0-t) | AUC(0-t) Ratio = Exp { [loge([14C]-GSK2269557 AUC(0-t)] - [loge(Total radioactivity AUC(0-t)] } Per subject for radiolabelled IV dose. |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.
- The 10 PK parameters AUC(0-t), AUC(0-24), AUC(0-inf), AUCex, Cmax, tmax, t1/2, CL, Vdss and Vc will be derived from phoenix and sent to S&P. The radiometric IV and oral dose will be calculated by Covance and sent to S&P. Additional parameters will be derived by S&P including CLr, ML(iv), ML(po), Fg, EH, Fabs, F and the treatment ratios

 Table 2
 Derived Urine and Faeces Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| Ae[urine] | Total radioactivity recovered in the urine (Ae[urine]) calculated for each collection interval |
| | per subject and treatment period as: |
| | Activinal (consentration in unine complex) |
| | Ae[urine]= (concentration in urine sample x collected sample weight) |
| | for each urine collection interval, eg 0-6, 6-24, 24-48, etc. |
| Cumulative<br>Ae[urine] | Cumulative total radioactivity recovered in the urine (Cumulative Ae[urine]) calculated for each cumulative collection interval per subject and treatment period as: |
| / to[uiiio] | , |
| | Cumulative Ae[urine]= summation of Ae[urine] |
| | for each urine collection within the cumulative urine collection interval, eg 0-24, 0-48, etc. |
| Fe%[urine] | % of total dose excreted as total radioactivity (Fe%[urine]) for each collection interval per |
| | subject and treatment period, will be estimated as: |
| | Fe%[urine]=(Ae[urine]) for each collection period)/Dose*100. |
| | Where the dose is the radiolabelled [14C]-GSK2269557, that is in period 1 radiometric iv |
| | dose, in period 2 radiometric oral dose |
| Cumulative | Cumulative % of total dose excreted as total radioactivity (Cumulative Fe%[urine]) for each |
| Fe%[urine] | cumulative collection interval per subject and treatment period, will be estimated as: |
| | Cumulative Fe%[urine]=summation of Fe%[urine] |
| | for each urine collection within the cumulative urine collection interval, eg 0-24, 0-48, etc. |

| Parameter | Parameter Description |
|---|---|
| Ae[faeces] | Total radioactivity recovered in the faeces (Ae[faeces]) calculated for each collection interval per subject and treatment period as |
| | Ae[faeces] = (concentration in faecal homogenate aliquot analysed x weight of homogenate aliquot analysed) x (total homogenate weight / collected sample weight) for each faecal collection interval, eg 0-24, 24-48, etc |
| Cumulative<br>Ae[faeces] | Cumulative total radioactivity recovered in the faeces (Cumulative Ae[faeces]) calculated for each cumulative collection interval per subject and treatment period as |
| | Cumulative Ae[faeces]= summation of Ae[faeces] for each faecal collection within the cumulative faecal collection interval, eg 0-24, 0-48, etc |
| Fe%[faeces] | % of total dose excreted as total radioactivity (Fe%[faeces]) for each collection interval per subject and treatment period will be estimated as: |
| | Fe%[faeces] =(Ae[faeces] for each collection period)/Dose*100. |
| | Where the dose is the radiolabelled [14C]-GSK2269557, that is in period 1 radiometric iv dose, in period 2 radiometric oral dose |
| Cumulative<br>Fe%[ faeces] | Cumulative % of total dose excreted as total radioactivity (Cumulative Fe%[ faeces]) for each cumulative collection interval per subject and treatment period will be estimated as: Cumulative Fe%[faeces]=summation of Fe%[faeces] |
| | for each faecal collection within the cumulative faecal collection interval, eg 0-24, 0-48, etc. |
| Ae[total] | Total radioactivity recovered in total excretion (sum of urine and faecal excretion), Ae[total] will be estimates by collection interval for each subject and treatment period as: |
| | Ae[total]=Ae[urine]+ Ae[faeces] |
| Cumulative<br>Ae[total] | Total radioactivity recovered in total excretion (sum of urine and faecal excretion), cumulative Ae[total] will be estimates by cumulative collection interval per subject and treatment period as: |
| | Cumulative Ae[total]= summation of Ae[total] |
| | for each total excretion collection within the cumulative total excretion collection interval, eg 0-24, 0-48, etc |
| Fe%[total] | % of total dose excreted as total radioactivity (Fe%[ total]) for each collection period will be estimated for each subject and treatment period as: |
| | Fe%[total]= Fe%[urine]+ Fe%[faeces] |
| Cumulative<br>Fe%[total] | Cumulative % of total dose excreted as total radioactivity (Cumulative Fe%[ total]) for each cumulative collection period will be estimated for each subject and treatment period as: |
| | Cumulative Fe%[total]= Cumulative Fe%[urine]+ Cumulative Fe%[faeces] |
| | for each total excretion collection within the cumulative total excretion collection interval, eg 0-24, 0-48, etc |

## NOTES:

• Additional parameters may be included as required.

## 8.2. Primary Pharmacokinetic Analyses

## 8.2.1. Endpoint / Variables

## 8.2.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Standards for Pharmacokinetic)

#### 8.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated as described in Section 8.1.2.

## 8.2.2. Summary Measure

A primary objective is to determine total radioactivity (drug related material) in plasma following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled GSK2269557 dose) and a single oral dose of [14C]-GSK2269557. To assess this, the plasma PK parameters: AUC (0-inf), AUC (0-t), AUC (0-24), %AUCex, Cmax, tmax, t1/2 of total drug-related material (radioactivity) will be summarised and listed.

The additional primary objective is to determine the rate and extent of excretion of total radioactivity in urine and faeces and the total recovery of radioactivity following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C]-GSK2269557. To assess this, the PK parameters: Ae and Fe% will be summarised and listed for urine faeces and total (Urine + Faeces).

#### 8.2.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

#### 8.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.3. Secondary Pharmacokinetic Analyses

## 8.3.1. Endpoint / Variables

#### 8.3.1.1. Drug Concentration Measures

Refer to Appendix 4 Data Display Standards & Handling Conventions (Section 11.4.3 Reporting Standards for Pharmacokinetic)

#### 8.3.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated as described in Section 8.1.2.

#### 8.3.2. Summary Measure

A secondary objective is to determine parent GSK2269557 concentration in plasma following a single IV microtracer of [14C]-GSK2269557 (concomitant with an inhaled non-radiolabelled GSK2269557 dose) and a single oral dose of [14C]-GSK2269557. To assess this, the plasma PK parameters: AUC (0-inf), AUC (0-t), AUC (0-24), %AUCex, Cmax, tmax, t1/2 of parent GSK2269557 ([14C]-GSK2269557 and GSK2269557) will be summarised and listed and the volume (Vdss and Vc) and clearance of parent GSK2269557 ([14C]-GSK2269557) after IV dose only will be summarised and listed.

Another secondary objective is to estimate the absolute bioavailability of GSK2269557 following inhaled and oral administration. To assess this, the oral and inhaled bioavailability (F) will be summarised and listed.

To assess metabolism, the plasma PK parameters: ML(iv), ML(po),  $F_g$ ,  $E_H$ ,  $F_{abs}$  will be summarised and listed. To assess exposure and metabolite ratio in humans, the ratio of Parent GSK2269557/total radioactivity will be calculated for the plasma PK parameters: Cmax, AUC(0-t), AUC(0-24) and  $AUC(0-\infty)$ , results will be summarised, listed and statistical analyses will be conducted as described in Section 8.3.4.1. To assess renal clearance, the PK CLr will be summarised and listed if bioanalysis can quantify parent GSK2269557 in urine collection intervals (i.e. if Ae is quantifiable for collection intervals).

### 8.3.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 8.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9 List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.3.4.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

Parent GSK2269557/Total radioactivity ratio for Cmax, AUC(0-t), AUC(0-24) and AUC(0-∞)

#### **Model Specification**

NOTE: The description below describes the current thinking of how to analyse these endpoints. The

proposed models will be assessed, and if not appropriate alternative models could be used.

[¹⁴C]-GSK2269557/ Total radioactivity ratio for Cmax, AUC(0-t), AUC(0-24) and AUC(0-∞) - Period 1 IV Dose

Following sample analyses the Parent GSK2269557 for the IV dose is likely to be presented as [14C]-GSK2269557 depending on the method, this is in addition to the Parent GSK2269557 for the inhaled dose and the total radioactivity. Analysis has been described for the [14C]-GSK2269557 analyte however may be adapted if alternate sample analysis is conducted.

For each period, following loge-transformation of plasma pharmacokinetic parameters of [¹⁴C]-GSK2269557 (from period 1 IV dose) and total radioactivity (from period 1 IV dose), AUC(0-∞), AUC(0-24), AUC(0-t) and Cmax will be separately analysed using a mixed effects model fitting a fixed effect term for analytes ([¹⁴C]-GSK2269557 (from period 1 IV dose) and total radioactivity (from period 1 IV dose)) and a random effect for subject. The Kenward & Roger (KR) degrees of freedom approach will be used. Point estimates for the mean difference between the [¹⁴C]-GSK2269557 and total radioactivity analytes, and associated 95% confidence interval will be constructed using the residual variance.

GSK2269557/ Total radioactivity ratio for Cmax, AUC(0-t), AUC(0-24) and AUC(0-∞) - Period 2 oral dose Following sample analyses the Parent GSK2269557 will be presented as either GSK2269557 or [14C]-GSK2269557 depending on the method, in addition to total radioactivity. Analysis has been described for parent GSK2269557 analyte and should be adapted to the appropriate analyte as appropriate. For each period, following loge-transformation of plasma pharmacokinetic parameters of Parent GSK2269557 (from period 2 oral dose) and total radioactivity (from period 2 oral dose), AUC(0-∞), AUC(0-24), AUC(0-t) and Cmax will be separately analysed using a mixed effects model fitting a fixed effect term for analytes (Parent GSK2269557 (from period 2 oral dose) and total radioactivity (from period 2 oral dose)) and a random effect for subject. The Kenward & Roger (KR) degrees of freedom approach will be used. Point estimates for the mean difference between the Parent GSK2269557 and total radioactivity analytes, and associated 95% confidence interval will be constructed using the residual variance.

## **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Normality assumptions underlying the model used for analysis will be examined by obtaining a normal
  probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the
  normality assumption and constant variance assumption of the model respectively) to gain confidence
  that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data

#### **Model Results Presentation**

 Point estimates for the mean difference between the Parent GSK2269557 and total radioactivity analytes, and associated 95% confidence interval will be constructed using the residual variance. The point estimate and confidence interval will then be exponentially back-transformed to obtain point estimates and associated 95% confidence interval for the ratio Parent GSK2269557/total radioactivity. These will be presented in a tabular form.

#### Sensitivity Analyses

 Data will be reviewed and if there are deviation that may affect the PK results, sensitivity analyses may be conducted as appropriate which may include excluding individual time points or excluding individual subjects as appropriate.

## 9. EXPLORATORY ANALYSES

As outlined in the protocol, there is an exploratory endpoint of characterisation and quantification of metabolites in plasma, urine, faeces, and duodenal bile. These analytical investigations may be conducted by GSK PTS IVIVT and the results reported in a separate GSK PTS IVIVT report.

## 10. REFERENCES

Davis,B and Morris,T. Physiological Parameters in Laboratory Animals and Humans. Pharmaceutical ResearchVol10.No.7.1093-1095.1993.

PKOne and relevant information on Standards for the Transfer and Reporting of PK Data using HARP available within IDSL standards, 2008.

Protocol Deviation Management Plan for an open-label study in healthy male subjects, to determine the excretion balance and pharmacokinetics of [<sup>14</sup>C]-GSK2269557, administered as a single intravenous microtracer (concomitant with an inhaled non-radiolabelled dose) and a single oral dose, 2017

## 11. APPENDICES

## 11.1. Appendix 1: Protocol Deviation Management

- As detailed in Section 4.1, Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan and a listing and summary of important Protocol Deviations will be provided.
- A Per Protocol Population is not being defined for this study. However additional exploratory sensitivity summaries may be considered, if there are protocol deviations that may affect the primary PK endpoints. Any additional sensitivity summaries will be documented in the CSR.

## 11.2. Appendix 2: Schedule of Activities

## 11.2.1. Protocol Defined Schedule of Events

## **Schedule of activities for Treatment Period 1**

| Schedule of activities for Treatment Perio | Screening | | | Treatme | nt Perio | od 1 (IV | and inh | aled dos | ing) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Streeming | | | 110001110 | Da | | | area aos | ···s) | | |
| Procedure | | | 1 | | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| | -30 to -1 | -1 | Pre-<br>dose | Post- dose<br>0-16 h | 24 h | 48 h | 72 h | 96 h | 120 h | 144 h | 168 h |
| Admission to Unit | | X | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | |
| Discharge from Unit | | | | | | | | | | | X |
| Demographics | X | | | | | | | | | | |
| Full Physical Exam | X | | | | | | | | | | |
| Brief Physical Exam | | X | | | | | | | | | X |
| Inhaler training <sup>1</sup> | | X | | | | | | | | | |
| Medical/medication/drug/alcohol history | X | | | | | | | | | | |
| HIV, Hep B and Hep C screen | X | | | | | | | | | | |
| Alcohol and cotinine tests, and urine drugs of abuse <sup>2</sup> | X | X | | | | | | | | | |
| Laboratory safety tests | X | X | X | | X | | | | | | X |
| 12-lead ECG <sup>3</sup> | X | X | X | X | X | | | | | | X |
| Vital signs (HR and BP) <sup>3</sup> | X | X | X | X | X | | | | | | X |
| Inhaled dose | | | | X | | | | | | | |
| IV infusion | | | | $X^4$ | | | | | | | |
| Local tolerability assessment <sup>5</sup> | | | | X | X | X | | | | | |
| Blood samples for background radiation, total radioactivity, [14C]-GSK2269557 analysis and cold GSK2269557 analysis <sup>6</sup> | X <sup>7</sup> | $X^7$ | X <sup>7,8</sup> | X | X | X | X | X | | | X |
| Blood samples for metabolite profiling Urine collection <sup>10,11</sup> | | | $X^8$ | X <sup>9</sup> | | | | | | | |
| Urine collection <sup>10,11</sup> | | | X | X | X | X | X | X | X | X | X |
| Faecal collection <sup>12,13</sup> | | | $X^{13}$ | X | X | X | X | X | X | X | X |
| Entero-Test <sup>14</sup> | | | $\leftarrow$ | $\stackrel{=}{\longrightarrow}$ | | | | | | | |
| Meals <sup>15</sup> | | | | X | | | | | | | |

| | Screening Treatment Period 1 (IV and inhaled dosing) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day | | | | | | | | | | |
| Procedure | | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |
| | -30 to -1 | -1 | Pre-<br>dose | Post- dose<br>0–16 h | 24 h | 48 h | 72 h | 96 h | 120 h | 144 h | 168 h |
| AE/concomitant medication review <sup>16</sup> | | $\leftarrow$ | | | • | • | | | • | | $\longrightarrow$ |

- 1. Training conducted by reviewing the Patient Information Leaflet with the participant. Additional training may be conducted at the discretion of the investigator.
- 2. Breath test will be performed to check alcohol consumption. Both CO breath tests and urine cotinine tests will be performed to check smoking state.
- 3. Triplicate measurements will be taken at screening and pre-dose on Day 1; single measurements will be taken at 6 h post-dose on Day 1 and at all other time points. Mean of triplicate measurements to be used as baseline.
- 4. IV infusion to begin as soon as possible (but within 5 min) after the start of the inhaled dose.
- 5. Local tolerability assessment for injection site reactions will be performed immediately after the end of dosing on Day 1 at 6 and 12 h, and on Days 2 and 3.
- 6. Sampling times relative to the start of the IV infusion. Blood samples for total radioactivity, [14C]-GSK2269557 analysis and cold GSK2269557 analysis will be taken: pre-dose and at 0h (post inhalation and pre-IV infusion), at the end of infusion and at 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 168 h after the start of infusion.
- 7. Background radiation sample taken at screening, Day –1 and pre-dose only.
- 8. An additional pre-dose blood sample may be taken from 1 participant for preparation of a plasma shipment control (details provided in the SRM).
- 9. Blood samples for plasma metabolite profiling will be collected at 0.5 h and 4 h after the start of the IV infusion.
- 10. An aliquot from each urine collection will be taken for metabolic profiling (separate study).
- Sampling times relative to the start of the IV infusion. Urine will be collected at pre-dose, 0-6 h, 6-24 h then over 24 h collection periods as follows: 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h, 144-168 h.
- 12. An aliquot from each homogenised faecal collection will be taken for metabolic profiling (separate study).
- 13. Sampling times relative to the start of IV infusion The pre-dose faecal collection sample can be collected up to 24 h pre-dose. Afterward faeces will be collected over 24 h collection periods as follows: 0-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h, 144-168h.
- 14. Entero-Test string device will be swallowed at approximately 3.5 h pre-dose (start of inhaled dose) while participants are in a fasted state and the string removed at about 2.5 h post-dose on Day 1. At about 0.5 h post-dose (i.e. 2 hours before string withdrawal) a food cue will be used to stimulate gall bladder emptying).
- 15. Meal times are 30 min, 4 h and 10 h post dose on Day 1. On all other days, meals will be served at the standard times for the unit.
- 16. AEs and SAEs will be collected from the signing of the ICF until the follow-up visit. However, any SAEs related to study participation or a GSK concomitant medication will be recorded from the time a participant consents to participate in the study and until the final follow-up visit contact.

## Schedule of activities for treatment period ${\bf 2}$

| | Treatment Period 2 (Oral dosing) Day | | | | | | | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|
| n . | | | | | | | | | | | (7-14 days<br>post-last dose) <sup>2,3</sup> |
| Procedure | | | 1 <sup>1</sup> | 2 | 3 | 4 | 5 | 6 | 7 | 8 | |
| | -1 | Pre-dose | Post-dose<br>0-16 h | 24 h | 48 h | 72 h | 96 h | 120 h | 144 h | 168 h | |
| Admission to Unit | X | | | | | | | | | | |
| Discharge from Unit <sup>2,3</sup> | | | | | | | | | | X | |
| Drugs of abuse | X | | | | | | | | | | |
| Alcohol and cotinine tests <sup>4</sup> | X | | | | | | | | | | |
| Brief Physical Exam | | X | | | | | | | | | X |
| Laboratory safety tests | X | X | | X | | | | | | X | X |
| 12-lead ECG | X | X | X <sup>5</sup> | X | | | | | | X | X |
| Vital signs (HR and BP) | X | X | X <sup>5</sup> | X | | | | | | X | X |
| Oral dose | | | X | | | | | | | | |
| Blood samples for total radioactivity, [14C]-GSK2269557 analysis and cold GSK2269557 analysis | | X <sup>6</sup> | X | X | X | X | X | | | X | |
| Blood samples for metabolite profiling | | X | X <sup>7</sup> | X | | | | | | | |
| Urine collection <sup>8,9</sup> | | X | X | X | X | X | X | X | X | X | |
| Faecal collection <sup>10,11</sup> | | X <sup>11</sup> | X | X | X | X | X | X | X | X | X <sup>12</sup> |
| Meals <sup>13</sup> | | | X | | | | | | | | |
| AE/concomitant medication review <sup>14</sup> | < | | | | | | | | | | $\rightarrow$ |

- 1. There will be a washout of at least 14 days between dosing in treatment period 1 and 2.
- 2. If less than 1% of the dose is excreted in each 24 h period on Day 6 (120-144 h) and Day 7 (144-168 h) for a given participant, the participant may be discharged as early as Day 8 (after the LSC results are available), and no further samples (apart from for laboratory safety tests) will be collected. Follow-up procedures may be done at discharge and procedures scheduled for Day 8 and follow up will only be done once.
- 3. If excretion is higher than 1%, or if the results are inconclusive in each 24-h period on Day 6 (120-144 h) and Day 7 (144-168 h) for a given participant, that participant will remain at the unit, and urine and faecal collections will continue at 24-h intervals, for up to 7 days (until the morning of Day 15), until excretion is less than 1%. All remaining participants will be discharged from the unit on Day 15. Follow-up procedures may be done at discharge. In the unlikely event that excretion is still higher than 1% upon discharge on Day 15, participants will continue to collect faecal samples only, at home, at 24-h intervals. Samples collected at home will be returned to the clinic every 2-3 days.
- 4. Breath test will be performed to check alcohol consumption. Both CO breath tests and urine cotinine tests will be performed to check smoking state.
- 5. Vital signs and ECG will be taken 6 h post dose.
- 6. Sampling times relative to the oral dose. Blood samples for total radioactivity, [14C]-GSK2269557 analysis and cold GSK2269557 analysis will be taken: pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 h post-dose.
- 7. Blood samples for plasma metabolite profiling will be collected at 2 h and 6 h post-[14C]-GSK2269557oral dose.
- 8. An aliquot from each urine collection will be taken for metabolic profiling (separate study).
- 9. Urine will be collected at pre-dose, at 0-6 h, 6-24 h then over 24 h collection periods as follows: 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h, 144-168 h.
- 10. An aliquot from each faecal collection will be taken for metabolic profiling (separate study).
- 11. The pre-dose faecal sample can be collected up to 24 h pre-dose. Afterward faeces will be collected over 24 h collection periods as follows: 0-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h, 144-168 h.
- 12. If dose excretion is still higher than 1% after day 15 the participants will continue to collect faecal samples only, at home, at 24-h intervals until excretion is less than 1%.
- 13. Meal times are 4h and 10h post dose on Day 1. On all other days, meals will be served at the standard times for the unit.
- 14. AEs and SAEs will be collected from the signing of the ICF until the follow-up visit. However, any SAEs related to study participation or a GSK concomitant medication will be recorded from the time a participant consents to participate in the study and until the final follow-up visit contact.

# 11.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 11.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the start and/or stop time/date of the study treatment within the period (for period 1 the inhaled and IV dose, for period 2 the oral dose).

These treatment phases are already defined in the Time and Event table in Appendix 2 Schedule of Activities (Section 11.2).

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time < Date/Time ≤ Study Treatment Stop Date/Time |
| Post-Treatment | Date/Time > Study Treatment Stop Date /Time |

## 11.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### **Treatment Emergent Flag for Adverse Events** 11.3.2.

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date plus washout. |
| | • Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 14 days. |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period:</li> <li>Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date +14 days.</li> </ul> |

## NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment. Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

#### 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. **Reporting Process**

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : UK1SAL00175 |
| HARP Compound | : GSK2269557 |
| HARP Study | : mid206764 |
| Analysis Datasets | |

Analysis datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) standards. If the Study Data Standardization Plan (SDSP) exists for a study, ensure the CDISC versions are consistent.

#### **Generation of RTF Files**

RTF files will be generated for summary tables.

#### 11.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the pCRF.
- The reported precision from non pCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visi | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

## 11.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non- | PC WNL file (CSV format) for the non compartmental analysis by Clinical |
| Linear (WNL) File | Pharmacology Modelling and Simulation function will be created according to PKOne. |
| | Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary Statistics, Graphical | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| Plasma PK Parameter to be Derived by Programmer | The following PK parameters will be derived by the Programmer: CLr, ML(iv), ML(po), Fg, E <sub>H</sub> , F <sub>abs</sub> , F(Oral, (0-t)), F(Oral, (0- $\infty$ )), F(inhaled, (0-t)), F (inhaled, (0- $\infty$ )) and the Parent GSK2269557/ Total Radioactivity ratio for Cmax, AUC(0-t), AUC(0-24) and AUC(0- $\infty$ ). note: Parent GSK2269557/ Total Radioactivity ratios will be either GSK2269557/ Total Radioactivity or [14C]-GSK2269557/ Total Radioactivity depending on the method of sample analyses and are of interest for the radiolabelled IV and oral dose. |
| Urine and Faeces PK Parameter to be Derived by Programmer | The following PK parameters will be derived by the Programmer: cumulative Ae, Fe% and cumulative Fe%. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to PKOne |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Triplicate measures of 12-lead ECG and vital signs (HR and BP) will be taken at screening and pre
  dose for period 1. The mean of the measurements will be calculated and used in any derivation of
  summary statistics but if listed all data will be presented.
- There are no other scheduled multiple measurements however, if multiple measurements are recorded at a given time point the following process will be followed:
  - [1] Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
  - [2] If there are two values within a time window (as per Section 11.2) the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
  - [3] Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 11.5.2. Study Population

## **Study Population**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
  - The year of the birth date will be captured in the pCRF

Age will then be derived as the integer value of [(DoB- date of Screening)/365.25]

• Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m) 2]

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as 1 day in period 1 and 1 day in period 2.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### **Study Population**

### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 11.5.3. Safety

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcF is machine read, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the pCRF, corrected QT intervals by Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

This imputation should be performed on the raw data before the conversion of units in CDISC studies to ensure correct imputation of missing data.

## 11.6. Appendix 6: Reporting Standards for Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as one who has completed all phases of the study including the last visit.</li> <li>If participants prematurely discontinue the study, additional replacement participants may be enrolled at the discretion of the sponsor and in consultation with the investigator</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| Liver<br>Chemistry<br>Stopping<br>Criteria | <ul> <li>Study treatment will be stopped for a subject if the following liver chemistry stopping criteria is met: <ul> <li>ALT ≥ 3 x ULN; or</li> <li>ALT ≥ 3 X ULN and total bilirubin ≥ 2 x ULN (&gt; 35% direct bilirubin); or</li> <li>ALT ≥ 3 x ULN and INR &gt; 1.5 (INR is not a Protocol requirement)</li> </ul> </li> <li>Note: Refer to Appendix 4 of Protocol for details of the required assessments if a subject meets the above criteria.</li> </ul> |
| QTc<br>Stopping<br>Criteria | A subject who meets either bulleted criterion below will be withdrawn from the study: |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The pCRF allows for the possibility of partial dates (i.e., only month and/or year) to be recorded for AE start and end dates; that is, the day or the month of the date may be missing.</li> <li>Any fully or partially missing dates for adverse events will be raised to data management for resolution before DBR.</li> </ul> |
| Element | Reporting Detail | | | | | |
|---|---|--|--|--|--|--|
| | <ul> <li>If fully or partially missing dates are available following DBF, the following conventions<br/>will be applied for calculating the time to onset and the duration of the event:<br/>Partially Missing Dates:</li> </ul> | | | | | |
| | Missing Start Day: First of the month will be used unless this is before the start<br>date of study treatment; in this case the latest study treatment start date will be<br>used and hence the event is considered On-treatment as per Appendix 3 Study<br>Phases and Treatment Emergent Adverse Events. | | | | | |
| | Missing Start Month: January will be used unless this is before the start date of study treatment; in this case the month of the latest study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3 Study Phases and Treatment Emergent Adverse Events. | | | | | |
| | <ul> <li>Missing Start Year: Current year will be used unless this is before the start date of<br/>study treatment; in this case the year of the latest study treatment start date will be<br/>used and hence the event is considered On-treatment as per Appendix 3 Study<br/>Phases and Treatment Emergent Adverse Events.</li> </ul> | | | | | |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the latest study treatment stop date will be<br/>used.</li> </ul> | | | | | |
| | <ul> <li>Missing Stop Month: December will be used, unless this is after the stop date of<br/>study treatment; in this case the latest month of study treatment stop date will be<br/>used.</li> </ul> | | | | | |
| | <ul> <li>Missing Stop Year: Current year will be used, unless this is after the stop date of<br/>study treatment; in this case the latest year of study treatment stop date will be<br/>used.</li> </ul> | | | | | |
| | Fully Missing Dates: Completely missing start or end dates will remain missing, with no imputation applied. | | | | | |
| | Consequently, time to onset and duration of such events will be missing. | | | | | |
| Concomitant<br>Medications/ | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed<br/>using the following convention:</li> </ul> | | | | | |
| Medical<br>History | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be<br/>used for the month</li> </ul> | | | | | |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent<br/>on the month and year) and 'Dec' will be used for the month.</li> </ul> | | | | | |
| | The recorded partial date will be displayed in listings. | | | | | |

# 11.7. Appendix 7: Values of Potential Clinical Importance

# 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Haematocrit | Ratio of 1 | Male | | 0.54 |
| Haematocht | Ratio of 1 | $\Delta$ from BL | ↓0.075 | |
| Haamadahin | g/L | Male | | 180 |
| Haemoglobin | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | | | 1.3 x ULN |
| Creatinine | mmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | ≤ 450 |
| Absolute PR Interval | msec | < 120 | < 220 |
| Absolute QRS Interval | msec | | ≤ 120 |
| Absolute Ventricular rate | beats/min | <35 | >100 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

# 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|--------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 90 | ≤ 140 |
| Diastolic Blood Pressure | mmHg | ≥ 40 | ≤ 90 |
| Heart Rate | bpm | ≥ 40 | ≤ 90 |
| Respiration rate | breaths/min | ≥ 8 | ≤ 20 |
| Oral Temperature | °C | ≥ 35.5 | ≤ 37.8 |

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|----------|
| (Change from Baseline) | | Decrease | Increase |
| Systolic Blood Pressure | mmHg | ≥ 40 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 20 | ≥ 20 |
| Heart Rate | bpm | ≥ 30 | ≥ 30 |

# 11.8. Appendix 8: Abbreviations & Trade Marks

# 11.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| pCRF | Paper Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |

| Abbreviation | Description |
|--------------|------------------------------|
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

# 11.8.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

### 11.9. Appendix 9: List of Data Displays

### 11.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.11 | N/A |
| Pharmacokinetic | 2.1 to 2.20 | 2.1 to 2.17 |
| Safety | 3.1 to 3.11 | N/A |
| Section | List | ings |
| ICH Listings | 1 to 30 | |
| Other Listings | 31 to 46 | |

### 11.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|-------|---------|
| Study Population | N/A | N/A | N/A |
| Pharmacokinetic | N/A | N/A | N/A |
| Safety | N/A | N/A | SAFE_L1 |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 11.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 11.9.4. Study Population Tables

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | • |
| 1.1. | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch | ICH E3 | SAC |
| 1.4. | APE | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoco | ol Deviation | | | | • |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| 1.6. | Safety | IE2 | Summary of Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | tion Analysed | | | | |
| 1.7. | Safety | SP1 | Summary of Study Populations | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.8. | Safety | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.9. | Safety | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.10. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Prior ar | Prior and Concomitant Medications | | | | |
| 1.11. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 | SAC |

### 11.9.5. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | | | | | |
| 2.1. | PK | PK01 | Summary of Plasma Total Radioactivity Concentrations by Treatment and Time | Include un transformed concentrations | SAC |
| 2.2. | PK | Refer to<br>Programming<br>Notes | Summary of Log Transformed Plasma Total Radioactivity Concentrations by Treatment and Time | Include log transformed concentrations use standard macro for sumstatsinrows for log transformed variable, present similar to example shell PK01 but present geometric mean and SD (Log) rather than mean and SD respectively. | SAC |
| 2.3. | PK | PK03 | Summary of Derived Plasma Total Radioactivity PK Parameters by Treatment | Include columns for parameter, period, treatment, N, n, arithmetic mean, 95% CI of arithmetic mean, standard deviation (SD), median, minimum and maximum. | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.4. | PK | PK05 | Summary of Log-Transformed Derived Plasma Total Radioactivity PK Parameters by Treatment | Include columns for parameter, period, treatment, N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data, median, minimum, maximum and between subject geometric coefficient of variation (CVb (%)). Refer to Section 11.4.3 for parameters that should be log transformed refer to gsk2269557/pii115119/part_a/drivers/t_pk_sum_log (Table 4.3) | SAC |
| 2.5. | PK | PK01 | Summary of Plasma [14C]-GSK2269557 Concentrations by Treatment and Time | Include un transformed concentrations | SAC |
| 2.6. | PK | Refer to<br>Programming<br>Notes | Summary of Log Transformed Plasma [14C]-GSK2269557<br>Concentrations by Treatment and Time | Include log transformed concentrations use standard macro for sumstatsinrows for log transformed variable, present similar to example shell PK01 but present geometric mean and SD (Log) rather than mean and SD respectively. | SAC |
| 2.7. | PK | PK03 | Summary of Derived Plasma [14C]-GSK2269557 PK Parameters by Treatment | Include columns for parameter, period, treatment, N, n, arithmetic mean, 95% CI of arithmetic mean, standard deviation (SD), median, minimum and maximum. In addition to standard [14C]-GSK2269557 pk parameters include Clearance (CL(iv) and CLr) and volume (Vdss and Vc). | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | Include columns for parameter, period, treatment, N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data, median, minimum, maximum and between subject geometric coefficient of variation (CVb (%)). | |
| 2.8. | PK | PK05 | Summary of Log-Transformed Derived Plasma [14C]-GSK2269557 PK Parameters by Treatment | Refer to Section 11.4.3 for parameters that should be log transformed. In addition to standard [14C]-GSK2269557 pk parameters include Clearance (CL(iv) and CLr) and volume (Vdss and Vc). | SAC |
| | | | | gsk2269557/pii115119/part_a/drivers/t_<br>pk_sum_log (Table 4.3) | |
| 2.9. | PK | PK01 | Summary of Plasma GSK2269557 Concentrations by Treatment and Time | Include un transformed concentrations | SAC |
| 2.10. | PK | Refer to<br>Programming<br>Notes | Summary of Log Transformed Plasma GSK2269557 Concentrations by Treatment and Time | Include log transformed concentrations use standard macro for sumstatsinrows for log transformed variable, present similar to example shell PK01 but present geometric mean and SD (Log) rather than mean and SD respectively. | SAC |
| 2.11. | PK | PK03 | Summary of Derived Plasma GSK2269557 PK Parameters by Treatment | Include columns for parameter, period, treatment, N, n, arithmetic mean, 95% CI of arithmetic mean, standard deviation (SD), median, minimum and maximum. | SAC |

| Pharma | cokinetic: Table | s | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.12. | PK | PK05 | Summary of Log-Transformed Derived Plasma GSK2269557 PK Parameters by Treatment | Include columns for parameter, period, treatment, N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data, median, minimum, maximum and between subject geometric coefficient of variation (CVb (%)). Refer to Section 11.4.3 for parameters that should be log transformed refer to gsk2269557/pii115119/part_a/drivers/t_pk_sum_log (Table 4.3) | SAC |
| 2.13. | PK | PK06 | Summary of Oral and Inhaled Absolute Bioavailability | Refer to Section 11.4.3 for parameters that should be log transformed. Include PK Parameters: Inhaled F (0-∞), Inhaled F (0-t), Oral F (0-∞) and Oral F (0-t), Dose(Inhaled), Dose(iv) and Dose(Oral). Note: Dose(iv) and Dose(Oral) is radiometric dose, Dose(Inhaled) is nominal | SAC |
| 2.14. | PK | PK06 | Summary of Metabolic, Hepatic Extraction and Absorption Parameters | Refer to Section 11.4.3 for parameters that should be log transformed. Include PK Parameters: ML(iv), ML(po), F <sub>g</sub> , E <sub>H</sub> and F <sub>abs</sub> | SAC |

| Pharma | cokinetic: Table | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.15. | PK | [Non-Standard]<br>Refer to<br>Programming<br>notes | Summary of Parent GSK2269557/Total Radioactivity Ratio for Cmax, AUC(0-24), AUC(0-∞) and AUC(0-t) | Include columns for: period, parent GSK2269557/total radioactivity ratio (GSK2269557/total radioactivity or 14C-GSK2269557/ total radioactivity), parameter (Cmax, AUC(0-24), AUC(0-∞) or AUC(0-t)), geometric mean for ratio, SD(log), 95% CI, median, minimum, maximum and between subject geometric coefficient of variation (CVb (%)). | SAC |
| 2.16. | PK | [Non-Standard]<br>Refer to<br>Programming<br>notes | Summary of Statistical Analyses for Parent GSK2269557/Total Radioactivity Ratio for Cmax, AUC(0-24), AUC(0-∞) and AUC(0-t) | Include columns for: period, parent GSK2269557/total radioactivity ratio (GSK2269557/total radioactivity or 14C-GSK2269557/ total radioactivity), parameter (Cmax, AUC(0-24), AUC(0-∞) or AUC(0-t)), estimate for ratio, SD(log) and 95% CI | SAC |
| Urine/F | aeces | | | | |
| 2.17. | PK | PK02 | Summary of Urinary and Faecal –Total Radioactivity Pharmacokinetic Parameters (Amount Excreted) by Treatment and Time | Include Ae(urine), Ae(faeces) and Ae(total). | SAC |
| 2.18. | PK | PK02 | Summary of Urinary and Faecal –Total Radioactivity Pharmacokinetic Parameters (Cumulative Amount Excreted) by Treatment and Time | Include cumulative Ae(urine), Cumulative Ae(faeces) and Cumulative Ae(total). | SAC |
| 2.19. | PK | PK02 | Summary of Urinary and Faecal –Total Radioactivity Pharmacokinetic Parameters (% of Dose Excreted) by Treatment and Time | Include Fe%(urine), Fe%(faeces) and Fe%(total). | SAC |
| 2.20. | PK | PK02 | Summary of Urinary and Faecal –Total Radioactivity Pharmacokinetic Parameters (Cumulative % of Dose Excreted) by Treatment and Time | Include cumulative Fe%(urine), Cumulative Fe%(faeces) and Cumulative Fe%(total). | SAC |

# 11.9.6. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | | | | | |
| | | | | Linear and log plot on same page. Separate page per treatment. N (likely 6) lines for each treatment with legend to identify subjects | |
| 2.1. | PK | PK16a | Individual Subject Plasma Total Radioactivity-time Plot (Linear and Semi-log) by Treatment | Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote | SAC |
| | | | | refer to<br>GSK961081/mid201003/final/f_pk_21<br>(Table 2.1) | |
| 2.2. | PK | PK19 | Arithmetic Mean (+SD) Plasma Total Radioactivity-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote | SAC |
| | | | refer to GSK961081/ mid201003/ final/<br>f_pk_22 (Table 2.2) | | |
| 2.3. | PK | PK PK20 Median (Range) Plasma Total Radioactivity-time Plot (Linear and Semi-log) by Treatment | | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote | SAC |
| | | | refer to GSK961081/ mid201003/ final/<br>f_pk_23 (Table 2.3) | | |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.4. | PK | PK16a | Individual Subject Plasma [14C]-GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. N (likely 6) lines for each treatment with legend to identify subjects Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/mid201003/final/f_pk_21 | SAC |
| 2.5. | РК | PK19 | Arithmetic Mean (+SD) Plasma [14C]-GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/ mid201003/ final/ f_pk_22 | SAC |
| 2.6. | PK | PK20 | Median (Range) Plasma [14C]-GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/ mid201003/ final/ f_pk_23 | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.7. | PK | PK16a | Individual Subject Plasma GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. N (likely 6) lines for each treatment with legend to identify subjects Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/mid201003/final/f_pk_21 | SAC |
| 2.8. | PK | PK19 | Arithmetic Mean (+SD) Plasma GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/ mid201003/ final/ f_pk_22 | SAC |
| 2.9. | PK | PK20 | Median (Range) Plasma GSK2269557 Concentration-time Plot (Linear and Semi-log) by Treatment | Linear and log plot on same page. Separate page per treatment. Time = Planned time post dose (h) Include the LLOQ as a reference line and footnote refer to GSK961081/ mid201003/ final/ f_pk_23 | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Urine ar | nd Faeces | | | | |
| 2.10. | PK | PK_F4 | Individual Subject Absolute –Total Radioactivity Recovered (Amount Excreted) for Urine, Faeces and Total Excretion by Time and Treatment | Ae(urine), Ae(faeces), Ae(total). Linear scale only. Separate page per subject and treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/ f_pk_210 | SAC |
| 2.11. | PK | PK_F5 | Arithmetic Mean Absolute –Total Radioactivity Recovered (Amount Excreted) for Urine, Faeces and Total Excretion by Time and Treatment | Ae(urine), Ae(faeces), Ae(total). Linear scale only. Separate page per Treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/ f_pk_212 | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.12. | PK | PK_F4 | Individual Subject Cumulative –Total Radioactivity Recovered (Cumulative Amount Excreted) for Urine, Faeces and Total Excretion by Time and Treatment | Cumulative Ae(urine), Cumulative Ae(faeces), Cumulative Ae(total). Linear scale only. Separate page per subject and treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/f_pk_210 | SAC |
| 2.13. | PK | PK_F5 | Arithmetic Mean Cumulative –Total Radioactivity Recovered (Cumulative Amount Excreted) for Urine, Faeces and Total Excretion by Time and Treatment | Cumulative Ae(urine), Cumulative Ae(faeces), Cumulative Ae(total). Linear scale only. Separate page per Treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/f_pk_212 | SAC |

| Pharmad | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.14. | PK | PK_F4 | Individual Subject Absolute –Total Radioactivity Recovered (% of Dose) for Urine, Faeces and Total Excretion by Time and Treatment | Fe%(urine), Fe%(faeces), Fe%(total). Linear scale only. Separate page per subject and treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/ f_pk_210 | SAC |
| 2.15. | PK | PK_F5 | Arithmetic Mean Absolute –Total Radioactivity Recovered (% of Dose) for Urine, Faeces and Total Excretion by Time and Treatment | Fe%(urine), Fe%(faeces), Fe%(total). Linear scale only. Separate page per Treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/ f_pk_212 | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.16. | PK | PK_F4 | Individual Subject Cumulative –Total Radioactivity Recovered (Cumulative % of Dose) for Urine, Faeces and Total Excretion by Time and Treatment | Cumulative Fe%(urine), Cumulative Fe%(faeces), Cumulative Fe%(total). Linear scale only. Separate page per subject and treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/ f_pk_210 | SAC |
| 2.17. | PK | PK_F5 | Arithmetic Mean Cumulative –Total Radioactivity Recovered (Cumulative % of Dose) for Urine, Faeces and Total Excretion by Time and Treatment | Cumulative Fe%(urine), Cumulative Fe%(faeces), Cumulative Fe%(total). Linear scale only. Separate page per Treatment. 3 lines per plot with legend to identify Urine Faeces and Total Excretion Time = actual mid-point of collection post dose (h). refer to GSK961081/ mid201003/ final/f_pk_212 | SAC |

# 11.9.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Adverse | Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | Safety | AE1CP | Summary All Drug-Related Adverse Events | ICH E3 | SAC |
| Serious | and Other Signi | ficant Adverse Ever | nts | | |
| 3.3. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.4. | Safety | AE1CP | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | IDSL | SAC |
| Laborat | ory: Chemistry | | | | |
| 3.5. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC |
| Laborat | ory: Hematology | | | | |
| 3.6. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
| Laborat | Laboratory: Urinalysis | | | | |
| 3.7. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 | SAC |
| Laborat | ory: Hepatobiliai | y (Liver) | | | |
| 3.8. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |

| Safety: 7 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | |
| 3.9. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.10. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| Vital Sig | Vital Signs | | | | |
| 3.11. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |

# 11.9.8. ICH Listings

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | 1 |
| 1. | APE | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | APE | ES9 | Listing of Subjects Who Were Rescreened | | SAC |
| 3. | Safety | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 4. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3. | SAC |
| 5. | Safety | CP_TA2 | Listing of Planned and Actual Treatments | IDSL<br>non randomised study so do not say<br>"randomised" use "Planned" instead | SAC |
| Protoco | l Deviations | | | | |
| 6. | Safety | DV2A | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Populat | ions Analysed | | | · | |
| 8. | APE | SP3a | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demogr | aphic and Basel | ine Characteristics | | • | |
| 9. | Safety | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | Safety | DM10 | Listing of Race | ICH E3 | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Prior ar | nd Concomitant I | Medications | | | |
| 11. | Safety | CP_CM4 | Listing of Concomitant Medications | IDSL | SAC |
| Exposu | re and Treatmen | t Compliance | | | • |
| 12. | Safety | EX4 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | | • |
| 13. | Safety | AE9CP | Listing of All Adverse Events | ICH E3 | SAC |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | and Other Signi | ficant Adverse Eve | nts | | |
| 16. | Safety | AE9CPa | Listing of Serious Adverse Events | ICH E3 Include fatal and non fatal | SAC |
| 17. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 18. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 Include fatal and non fatal | SAC |
| Hepato | biliary (Liver) | | | | |
| 19. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 20. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| All Labo | All Laboratory | | | | |
| 21. | Safety | LB6 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 22. | Safety | LB6 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 23. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 24. | Safety | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| ECG | | | | | |
| 25. | Safety | CP_EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 26. | Safety | CP_EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 27. | Safety | CP_EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| 28. | Safety | CP_EG6 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital Sig | gns | | | | |
| 29. | Safety | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| 30. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL | SAC |

# 11.9.9. Non-ICH Listings

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Plasma | PK | | | | |
| 31. | PK | PK08 | Listing of Plasma Total Radioactivity-Time Data | | SAC |
| 32. | PK | PK14 | Listing of Derived Plasma Total Radioactivity Pharmacokinetic Parameters | | SAC |
| 33. | PK | PK08 | Listing of Plasma [14C]-GSK2269557 Concentration-Time Data | | SAC |
| 34. | PK | PK14 | Listing of Derived Plasma [14C]-GSK2269557 Pharmacokinetic Parameters | In addition to standard [14C]-GSK2269557 pk parameters include Clearance (CL(iv) and CLr) and volume (Vdss and Vc). | SAC |
| 35. | PK | PK08 | Listing of Plasma GSK2269557 Concentration-Time Data | | SAC |
| 36. | PK | PK14 | Listing of Derived Plasma GSK2269557 Pharmacokinetic Parameters | | SAC |
| 37. | PK | PK14 | Listing of Oral and Inhaled Absolute Bioavailability | Include PK Parameters: Inhaled F (0-∞), Inhaled F (0-t), Oral F (0-∞) and Oral F (0-t), Dose(Inhaled), Dose(iv) and Dose(Oral). Note: Dose(iv) and Dose(Oral) is radiometric | SAC |
| | | | | dose, Dose(Inhaled) is nominal | |
| 38. | PK | PK14 | Listing of Metabolic, Hepatic Extraction and Absorption Parameters | Include PK Parameters: ML(iv), ML(po), $F_g$ , $E_H$ and $F_{abs}$ | SAC |
| 39. | PK | PK15 | Listing of Individual Subject Parent GSK2269557/Total Radioactivity Ratio for Cmax, AUC(0-∞), AUC(0-24) and AUC(0-t) | | SAC |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Urine ar | Urine and Faeces PK | | | | |
| 40. | PK | [Non-Standard]<br>Refer to<br>programming<br>notes | Listing of Urinary and Faecal Total Radioactivity Parameters (Amount Excreted) by Time | Ae(urine), Ae(faeces), Ae(total) and cumulative Ae(urine), cumulative Ae(faeces), cumulative Ae(total) refer to GSK961081/ mid201003/ final/ I_pk_ae (listing 35) | SAC |
| 41. | PK | [Non-Standard]<br>Refer to<br>programming<br>notes | Listing of Urinary and Faecal Total Radioactivity Parameters (% Excreted) by Time | Fe%(urine), Fe%(faeces), Fe%(total) and cumulative Fe%(urine), cumulative Fe%(faeces), cumulative Fe%(total) refer to GSK961081/ mid201003/ final/ I_pk_fe (listing 36) | SAC |
| Liver M | onitoring | | | | |
| 42. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC |
| 43. | Safety | LIVER7 | Listing of Liver Biopsy Details | | SAC |
| 44. | Safety | LIVER8 | Listing of Liver Imaging Details | | SAC |
| 45. | Safety | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory Criteria Post-<br>Baseline | | SAC |
| Entero- | Test | | | | |
| 46. | Safety | [Non-Standard]<br>SAFE_L1 | Listing of Entero-Test Administration and Removal | | SAC |

# 11.10. Appendix 10: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request